CLINICAL TRIAL: NCT05553483
Title: Comparing the Effect of Laser Acupuncture Alone or Combined With Pranayama Exercise on Inflammatory Status/Markers in Children With Allergic Rhinitis
Brief Title: Effect of Laser Acupuncture Alone or Combined With Pranayama Exercise on Inflammation in Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003341
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pranayama and acupoint stimulation by laser (Experimental): for 6 weeks,This 30-children group will receive 2-session per-week laser stimulation to some selected acupoints and daily pranyama exercises (nearly every session will be one hour), the stimulated bilateral acupoints will be (LI 19, LI 20, ST2, and ST4. ST6, ST7, ST17, ST36, SI18, BL2, GB14, GV24 and EXHN5). Every acupoint will be stimulated with laser power of 100 mw that will be used on a spot area of 1 cm2 for 1 minute.
  this group will receive also pranayama session (applied daily, one hour approximately, for six weeks) will be (alternate nostril pranayama, diaphragmatic pranayama, rapid abdominal pranayama, Bhramari pranayama)
  Interventions: Other: pranayama plus acupoint stimulation by laser
- acupoint stimulation by laser (Active Comparator): for six weeks, This 30-children group will receive 2-session per-week laser stimulation to some selected acupoints. The stimulated bilateral points will be (LI 19, LI 20, ST2, and ST4. ST6, ST7, ST17, ST36, SI18, BL2, GB14, GV24 and EXHN5). Every acupoint will be stimulated with laser power of 100 mw that will be used on a spot area of 1 cm2 for 1 minute.
  Interventions: Other: acupoint stimulation by laser

INTERVENTIONS:
Other: pranayama plus acupoint stimulation by laser — This group will receive 2-session per-week laser stimulation (for six weeks) to some selected acupoints and daily pranyama exercises (nearly every session will be one hour), the stimulated bilateral acupoints will be (LI 19, LI 20, ST2, and ST4. ST6, ST7, ST17, ST36, SI18, BL2, GB14, GV24 and EXHN5). Every acupoint will be stimulated with laser power of 100 mw that will be used on a spot area of 1 cm2 for 1 minute.
  this group will receive also pranayama session (applied daily, one hour approximately, for six weeks) composed from (alternate nostril pranayama, diaphragmatic pranayama, rapid abdominal pranayama, Bhramari pranayama ).
  Arms: pranayama and acupoint stimulation by laser
Other: acupoint stimulation by laser — This group will receive 2-session per-week laser stimulation (for six weeks) to some selected acupoints. The stimulated bilateral acupoints will be (LI 19, LI 20, ST2, and ST4. ST6, ST7, ST17, ST36, SI18, BL2,GB14, GV24 and EXHN5). Every acupoint will be stimulated with laser power of 100 mw that will be used on a spot area of 1 cm2 for 1 minute.
  Arms: acupoint stimulation by laser

SUMMARY:
Allergic rhinitis (AR) represents one of the most common global health problems with seriously increasing incidence over the last decades.The goal of the treatment of rhinitis is to prevent or reduce the symptoms through reduction of the inflammation of affected tissues. Acupuncture and pranayama yoga exercises had reported a significant improvement in daily symptoms and an increase of symptom-free days in many studies enrolling patients.

DETAILED DESCRIPTION:
Sixty Egyptian children with allergic rhinitis, after randomization, will be divided to 2 groups; the first 30-children group will receive 2-session per-week laser stimulation for 6 weeks to some selected acupoints and daily pranyama exercises (nearly every session will be one hour, for six weeks), the second group will receive 2-session per-week laser stimulation for six weeks to some bilateral selected acupoints. the stimulated points will be (LI 19, LI 20, ST2, and ST4. ST6, ST7, ST17, ST36, SI18, BL2, GB14, GV24 and EXHN5). Every acupoint will be stimulated with laser power of 100 mw that will be used on a spot area of 1 cm2 for 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis children
* physician-based diagnosis of allergic rhinitis

Exclusion Criteria:

* children with intellectual disabilities
* chest disease or heart disease or local congenital nose deformities
* participants received within-previous-six-months self-prescribed or by-therapist prescribed complementary therapies

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — from the governmental birth certificate, gender is written in it
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
erothrocyte sidemention rate | It will be measured after 6 weeks
  it is a inflammatory marker in serum

SECONDARY OUTCOMES:
Immunoglobulin E | It will be measured after 6 weeks
  it is an antibody in the serum
interleukin 1-beta | It will be measured after 6 weeks
  it is a inflammatory marker in serum
C-reactive protein | It will be measured after 6 weeks
  it is a inflammatory marker in serum
total eosinophil count | It will be measured after 6 weeks
  it is a inflammatory marker in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt